CLINICAL TRIAL: NCT03455712
Title: Impact of a Patient Education Intervention on Maternal Knowledge of Gestational Weight Gain Recommendations
Brief Title: Impact of GWG Tool on Patient Knowledge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Allie Reid, Principal Investigator, MetroHealth Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB16-00295
Record Dates: First submitted 2018-02-27; First posted 2018-03-06 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Weight Gain; Pregnancy Related
Keywords: Pregnancy; Gestational weight gain; Weight gain; Patient education; Patient knowledge; Institute of Medicine
MeSH Terms: conditions — Weight Gain; Gestational Weight Gain

STUDY DESIGN:
Intervention Model Description: Subjects to be enrolled into the intervention and standard-of-care groups depending on their gestational age at the time of consent during the expected 2 month period of enrollment. Any subject who is between 6 weeks 0 days and 14 weeks 6 days of pregnancy at the time of consent and who has had no prior prenatal visits will be enrolled in the intervention group. Any subject who is between 15 weeks 0 days to 22 weeks 6 days of pregnancy at the time of consent and who has had at least one prior prenatal visit will be enrolled in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Subjects to receive the Gestational Weight Gain Card at enrollment in addition to standard prenatal care.
  Interventions: Behavioral: Gestational Weight Gain Card
- Standard-of-Care (No Intervention): No intervention to be delivered. Subjects to receive standard prenatal care.

INTERVENTIONS:
Behavioral: Gestational Weight Gain Card — The Gestational Weight Gain Card is designed to be an educational and weight gain tracking tool. Study subjects will be highly encouraged to use the GWG card to gain both important clinical information and to document weight measurements throughout their pregnancy.
  Arms: Intervention

SUMMARY:
Women with singleton pregnancies at one outpatient clinic to be recruited for controlled clinical trial. Over eight weeks, women 15 0/7--22 6/7 weeks' with at least one prior prenatal visit to be enrolled in the control group. Women 6 0/7--14 6/7 weeks' to be enrolled in the intervention group at their first prenatal visit and to receive a pregnancy-specific gestational weight gain card. Women to be encouraged to record their weight at each prenatal care visit. All women to complete a GWG knowledge--based questionnaire at 15 0/7-22 6/7 weeks'.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestation
* Primary prenatal care at MetroHealth Medical Center
* Planning to deliver at MetroHealth Medical Center

Exclusion Criteria:

* Any inclusion criteria not met
* Prior diagnosis of eating disorder
* Inadequate knowledge of English language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-06-27 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2017-09-07 (Actual)

PRIMARY OUTCOMES:
Pregnancy-specific topic/guideline questionnaire responses | Outcome assessed up to 23 weeks gestation
  Comparison of number of participants in control vs. intervention groups who correctly answer multiple choice and free response questions related to pregnancy-specific topics and guidelines following intervention.

SECONDARY OUTCOMES:
Pregnancy-specific topic/guideline questionnaire responses | Outcome assessed up to 23 weeks gestation
  Description of general patient population knowledge of pregnancy-specific topics and guidelines from number of participants who correctly answer multiple choice and free response questions related to pregnancy-specific topics and guidelines prior to intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Erica Berggren, MD, MSCR, Principal Investigator — Case Western Reserve University School of Medicine, MetroHealth Medical Center

IPD SHARING:
Plan to Share IPD: No